CLINICAL TRIAL: NCT06027892
Title: Two-fraction Versus Five-fraction Stereotactic Radiotherapy for Localized Low- and Favorable Intermediate-risk Prostate Cancer: SABR-Dual
Brief Title: Two-fraction Versus Five-fraction Stereotactic Radiotherapy for Localized Prostate Cancer
Acronym: SABR-Dual
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC-0199-22; MOH_2022-08-30_012007 (Registry Identifier: Israel Ministry of Health)
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-08

CONDITIONS: PROSTATE CANCER
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Two-fraction stereotactic radiotherapy (Experimental): Participants receive stereotactic ablative radiotherapy in two treatments to a dose of 27 Gy, with the options to boost a high-grade lesion to 30 Gy
  Interventions: Radiation: Two-fraction stereotactic radiotherapy
- Five-fraction stereotactic radiotherapy (Active Comparator): Participants receive stereotactic ablative radiotherapy in five treatments to a dose of 40 Gy, with the options to boost a high-grade lesion to 45 Gy
  Interventions: Radiation: Five-fraction stereotactic radiotherapy

INTERVENTIONS:
Radiation: Two-fraction stereotactic radiotherapy — Definitive prostate radiotherapy will be delivered to a dose biologically comparable to 40 Gy in 5 treatments, but in only 2 treatments
  Arms: Two-fraction stereotactic radiotherapy
Radiation: Five-fraction stereotactic radiotherapy — Definitive prostate radiotherapy will be delivered to a standard stereotactic dose of 40 Gy in 5 treatments
  Arms: Five-fraction stereotactic radiotherapy

SUMMARY:
The goal of this clinical trial is to compare two dose schedules of stereotactic radiation therapy in patients with localized prostate cancer. Historically, external beam radiation to treat localized prostate cancer was given in small treatments over a period of multiple weeks. Recent studies have shown that with newer technologies and better understanding of how prostate cancer responds to radiation, the same effective dose can be given in as few as 5 treatments. This study is comparing this newer standard course of 5 treatments with an even shorter course of just 2 treatments. The dose for the 2 treatments is based on a form of internal radiation called brachytherapy, but in this study, that dose will be given using external radiation, without the need for invasive procedures.

In order to make sure that the radiation therapy is given in a way that minimizes the risk of side effects to the surrounding organs, including the rectum and bladder, prior to radiation a hydrogel material will be inserted behind the prostate in order to distance the rectum further from the prostate gland, and small gold markers will be inserted into the prostate to decrease any possible movement during treatment.

The main questions are whether 2-treatment radiation is tolerated as well and is as effective at treating prostate cancer, compared to the standard 5-treatment course of radiation.

DETAILED DESCRIPTION:
Following publication of multiple prospective clinical trials demonstrating the biochemical progression free survival (bPFS) benefits of high dose radiation for the curative treatment of localized prostate cancer, typical external beam radiotherapy (EBRT) courses ranged from 38-45 daily fractions delivered over 7.5-9 weeks. Over the past two decades, monumental advances in EBRT have been achieved, allowing significant shortening of the standard radiotherapy course. With diagnostic, imaging, and technological developments, the ability to deliver higher doses per fraction further expanded and an improved radiobiologic understanding of the response of prostate adenocarcinoma revealed that ultrahypofractionated regimen could take advantage of the comparatively low a/b ratio of prostate cancer cells. As a result of these two streams of development, stereotactic ablative radiation therapy (SABR) emerged as an accepted standard of care for definitive treatment in the low- and favorable intermediate-risk settings.

At both the individual and systems levels, efficient delivery of patient care and prudent utilization of medical resources is at the forefront. Given the ubiquity of prostate cancer and high volumes of patients in treatment centers across the globe, there remains meaningful potential for substantial improvements in patient throughput and cost of care. Presently, the shortest treatment courses for low- and favorable intermediate-risk prostate cancer are radical prostatectomy and low-dose-rate (LDR) brachytherapy, which offer an excellent likelihood of cure but entail degrees of invasiveness that may not be appropriate, feasible, or desirable for all patients, and include additional costs associated with operating room facilities and anesthesia. Surgical patients typically require a brief inpatient hospital stay. A comparable radiation therapy treatment course could help address many of these concerns and offer effective and efficient patient care.

A strong and mature precedent for a two-fraction course of high dose radiation can be found in the realm of high-dose-rate (HDR) brachytherapy. Under anesthesia, a radioactive source is programmed to traverse catheters that have been transperineally inserted into the prostate in order to produce a desired dose deposit. bPFS rates range between 91%-97% in the modern literature. While attempts were made to deliver single-fraction HDR brachytherapy (typical dose of 19 Gy), trials resulted in inferior oncologic outcomes, and to date, standard HDR treatment courses are comprised of two-fraction definitive treatment or single-fraction combined with EBRT. Radiobiologically, based on the particularly low a/b of prostate cancer cells and unique cell cycling, there is suggestion that at least two fractions are necessary for complete tumor eradication.

There exists, to date, limited data on the safety and effectiveness of prostate SABR delivered in fewer than five fractions. A recent proof-of-concept study by Greco et al compared single-dose SABR of 24 Gy to 5 fractions of 9 Gy in favorable intermediate and unfavorable intermediate risk patients. The results demonstrated comparable four-year prostate specific antigen outcomes for favorable intermediate disease though inferior PFS for unfavorable intermediate disease. Objective and patient reported genitourinary and gastrointestinal toxicities were not significantly different, though one of the 15 patients in the single-fraction arm experienced delayed grade 3 urethral stenosis. Magli et al published acceptable 1-year toxicity outcomes for a novel three-fraction regimen of SABR for low- and favorable intermediate-risk patients, to a dose of 40 Gy. MRI based planning was utilized, gold fiducials and a hydrogel spacer were placed, and a catheter was inserted in the bladder for each fraction. They observed rates of 11.9% and 1.7% acute grade 2 and 3 urinary toxicity, respectively, and 8.5% acute grade 2 rectal toxicity, all of which resolved by 12 months. Alayed et al published safety and efficacy results of their prospective single-cohort study of low- and intermediate-risk patients undergoing a two-fraction SABR regimen to a dose of 26 Gy. On their sample of 30 patients, they reported no acute grade 3+ gastrointestinal or genitourinary toxicity, and one instance each in later follow up, comparable or even slightly better than that from five-fraction protocols.

Multiple questions remain regarding the potential role for and safety of delivering SABR in fewer than five fractions. These include optimal patient selection, ideal dose fractionation, proper techniques to assure necessary avoidance of surrounding normal tissue, and how to balance dose to organs at risk with the accepted requirement of a planning target volume (PTV) to account for inevitable setup uncertainty. Importantly, recent endoscopic reports reveal notably high rates of rectal ulceration after dose-escalated SABR, and placement of a hydrogel spacer has been demonstrated to significantly reduce this risk. Placement of a resorbable hydrogel spacer to displace the rectum away from the high dose region, allowing for a posterior safety margin to account for potential intra-fractional motion, instead of a rectal balloon, is essential for accomplishing rectal sparing while facilitating additional assurance regarding treatment accuracy.

In the context of modern dose escalation, and in lieu of a strong body of HDR-brachytherapy data supporting a two-fraction approach to ultra-high dose treatment with initial experiences of two-fraction SABR, direct comparison of a non-invasive and broadly generalizable two-fraction SABR regimen to the standard approach of five-fraction regimen is logical. Institutional studies have emerged in the recent years demonstrating evidence for safety of ultra-hypofractionated regimen in fewer than five fractions of SABR, and large-scale randomized data is much needed. Aided by the ability to achieve necessary rectal dose constraints through placement of a rectal hydrogel, this approach may serve as an appropriate balance between minimizing the number of treatments necessary while allowing for delivery of the higher dose needed to optimize likelihood of cure.

ELIGIBILITY:
Inclusion:

* Male patients ≥18 years
* Diagnosis of low- or favorable intermediate-risk prostate adenocarcinoma

  * T1-T2c
  * Prostate specific antigen < 20
  * Gleason 6 or 7 (3+4)
  * Cannot had multiple intermediate-risk factors consistent with unfavorable intermediate risk disease
* Prostate gland < 60 cc (can include following cytoreductive androgen deprivation)
* International Prostate Symptom Score < 15 (unaided by a-adrenergic inhibitor or anticholinergic drugs)

Exclusion:

* Unfavorable intermediate-risk disease and above
* Chronic inflammatory bowel condition (IBD, Crohn's disease, Sarcoidosis, Rheumatic disease)
* Chronic immunosuppression
* Contraindications to hydrogel spacer placement
* Contraindications to a prostate MRI
* Any prior prostate cancer treatment
* Prior pelvic radiotherapy
* Previous transurethral resection of the prostate (TURP) within 12 months
* Hip prosthesis
* Prior use of therapeutic androgen deprivation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 562 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Biochemical Progression Free Survival | five-year
  Phoenix definition

SECONDARY OUTCOMES:
Freedom From Progression | five-year
  biochemical failure, clinical failure, death from any cause
Distant metastasis free survival | five-year
  Survival without development of distant metastatic disease
Prostate cancer specific survival | five-year
  Survival with cause of death or censoring without residual or recurrent prostate cancer
Time to prostate specific antigen nadir (< 0.2) - Longitudinal response | five-year
  Biochemical prostate specific antigen response over time
Time to salvage treatment | five-year
  Time interval until need for salvage treatment for residual or recurrent disease
Physician-reported Genitourinary/Gastrointestinal toxicity | Every 3 months until 24 months
  Toxicity caused by the intervention as graded by the physician
Patient-reported Genitourinary/Gastrointestinal toxicity | Every 3 months until 24 months
  Toxicity caused by the intervention as graded by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Elisha T Fredman, MD, Principal Investigator — Davidoff Cancer Center, Rabin Medical Center
Locations (1):
- Davidoff Cancer Center, Rabin Medical Center, Petah Tikva, Israel, Israel

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data used in the results publication will be provided with participating researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Individual participant data and supporting information will be made upon request through final publication of the study results
Access Criteria: Access will be granted by the leading study PI upon request by participating researchers, based on the needs and length of time necessary.
URL: https://rabin-medical.org/

REFERENCES:
- [Background] Gharzai LA, Jiang R, Wallington D, Jones G, Birer S, Jairath N, Jaworski EM, McFarlane MR, Mahal BA, Nguyen PL, Sandler H, Morgan TM, Reichert ZR, Alumkal JJ, Mehra R, Kishan AU, Fizazi K, Halabi S, Schaeffer EM, Feng FY, Elliott D, Dess RT, Jackson WC, Schipper MJ, Spratt DE. Intermediate clinical endpoints for surrogacy in localised prostate cancer: an aggregate meta-analysis. Lancet Oncol. 2021 Mar;22(3):402-410. doi: 10.1016/S1470-2045(20)30730-0. PMID 33662287
- [Background] Abramowitz MC, Li T, Buyyounouski MK, Ross E, Uzzo RG, Pollack A, Horwitz EM. The Phoenix definition of biochemical failure predicts for overall survival in patients with prostate cancer. Cancer. 2008 Jan 1;112(1):55-60. doi: 10.1002/cncr.23139. PMID 17968996
- [Background] Marcello M, Denham JW, Kennedy A, Haworth A, Steigler A, Greer PB, Holloway LC, Dowling JA, Jameson MG, Roach D, Joseph DJ, Gulliford SL, Dearnaley DP, Sydes MR, Hall E, Ebert MA. Reduced Dose Posterior to Prostate Correlates With Increased PSA Progression in Voxel-Based Analysis of 3 Randomized Phase 3 Trials. Int J Radiat Oncol Biol Phys. 2020 Dec 1;108(5):1304-1318. doi: 10.1016/j.ijrobp.2020.07.030. Epub 2020 Jul 30. PMID 32739320
- [Background] Folkert MR, Zelefsky MJ, Hannan R, Desai NB, Lotan Y, Laine AM, Kim DWN, Neufeld SH, Hornberger B, Kollmeier MA, McBride S, Ahn C, Roehrborn C, Timmerman RD. A Multi-Institutional Phase 2 Trial of High-Dose SAbR for Prostate Cancer Using Rectal Spacer. Int J Radiat Oncol Biol Phys. 2021 Sep 1;111(1):101-109. doi: 10.1016/j.ijrobp.2021.03.025. Epub 2021 Mar 19. PMID 33753140
- [Background] Kim DW, Cho LC, Straka C, Christie A, Lotan Y, Pistenmaa D, Kavanagh BD, Nanda A, Kueplian P, Brindle J, Cooley S, Perkins A, Raben D, Xie XJ, Timmerman RD. Predictors of rectal tolerance observed in a dose-escalated phase 1-2 trial of stereotactic body radiation therapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2014 Jul 1;89(3):509-17. doi: 10.1016/j.ijrobp.2014.03.012. PMID 24929162
- [Background] Alayed Y, Cheung P, Chu W, Chung H, Davidson M, Ravi A, Helou J, Zhang L, Mamedov A, Commisso A, Commisso K, Loblaw A. Two StereoTactic ablative radiotherapy treatments for localized prostate cancer (2STAR): Results from a prospective clinical trial. Radiother Oncol. 2019 Jun;135:86-90. doi: 10.1016/j.radonc.2019.03.002. Epub 2019 Mar 19. PMID 31015175
- [Background] Magli A, Farneti A, Faiella A, Ferriero M, Landoni V, Giannarelli D, Moretti E, de Paula U, Gomellini S, Sanguineti G. Toxicity at 1 Year After Stereotactic Body Radiation Therapy in 3 Fractions for Localized Prostate Cancer. Int J Radiat Oncol Biol Phys. 2021 Sep 1;111(1):93-100. doi: 10.1016/j.ijrobp.2021.03.027. Epub 2021 Mar 19. PMID 33745951
- [Background] Greco C, Pares O, Pimentel N, Louro V, Santiago I, Vieira S, Stroom J, Mateus D, Soares A, Marques J, Freitas E, Coelho G, Seixas M, Lopez-Beltran A, Fuks Z. Safety and Efficacy of Virtual Prostatectomy With Single-Dose Radiotherapy in Patients With Intermediate-Risk Prostate Cancer: Results From the PROSINT Phase 2 Randomized Clinical Trial. JAMA Oncol. 2021 May 1;7(5):700-708. doi: 10.1001/jamaoncol.2021.0039. PMID 33704378
- [Background] Morton G, McGuffin M, Chung HT, Tseng CL, Helou J, Ravi A, Cheung P, Szumacher E, Liu S, Chu W, Zhang L, Mamedov A, Loblaw A. Prostate high dose-rate brachytherapy as monotherapy for low and intermediate risk prostate cancer: Efficacy results from a randomized phase II clinical trial of one fraction of 19 Gy or two fractions of 13.5 Gy. Radiother Oncol. 2020 May;146:90-96. doi: 10.1016/j.radonc.2020.02.009. Epub 2020 Mar 5. PMID 32146259
- [Background] Viani GA, Arruda CV, Assis Pellizzon AC, De Fendi LI. HDR brachytherapy as monotherapy for prostate cancer: A systematic review with meta-analysis. Brachytherapy. 2021 Mar-Apr;20(2):307-314. doi: 10.1016/j.brachy.2020.10.009. Epub 2021 Jan 15. PMID 33461894
- [Background] Pickles T, Morris WJ, Kattan MW, Yu C, Keyes M. Comparative 5-year outcomes of brachytherapy and surgery for prostate cancer. Brachytherapy. 2011 Jan-Feb;10(1):9-14. doi: 10.1016/j.brachy.2009.12.004. PMID 20605535
- [Background] Hoffman KE, Penson DF, Zhao Z, Huang LC, Conwill R, Laviana AA, Joyce DD, Luckenbaugh AN, Goodman M, Hamilton AS, Wu XC, Paddock LE, Stroup A, Cooperberg MR, Hashibe M, O'Neil BB, Kaplan SH, Greenfield S, Koyama T, Barocas DA. Patient-Reported Outcomes Through 5 Years for Active Surveillance, Surgery, Brachytherapy, or External Beam Radiation With or Without Androgen Deprivation Therapy for Localized Prostate Cancer. JAMA. 2020 Jan 14;323(2):149-163. doi: 10.1001/jama.2019.20675. PMID 31935027
- [Background] Jackson WC, Silva J, Hartman HE, Dess RT, Kishan AU, Beeler WH, Gharzai LA, Jaworski EM, Mehra R, Hearn JWD, Morgan TM, Salami SS, Cooperberg MR, Mahal BA, Soni PD, Kaffenberger S, Nguyen PL, Desai N, Feng FY, Zumsteg ZS, Spratt DE. Stereotactic Body Radiation Therapy for Localized Prostate Cancer: A Systematic Review and Meta-Analysis of Over 6,000 Patients Treated On Prospective Studies. Int J Radiat Oncol Biol Phys. 2019 Jul 15;104(4):778-789. doi: 10.1016/j.ijrobp.2019.03.051. Epub 2019 Apr 6. PMID 30959121
- [Background] Lee WR, Dignam JJ, Amin MB, Bruner DW, Low D, Swanson GP, Shah AB, D'Souza DP, Michalski JM, Dayes IS, Seaward SA, Hall WA, Nguyen PL, Pisansky TM, Faria SL, Chen Y, Koontz BF, Paulus R, Sandler HM. Randomized Phase III Noninferiority Study Comparing Two Radiotherapy Fractionation Schedules in Patients With Low-Risk Prostate Cancer. J Clin Oncol. 2016 Jul 10;34(20):2325-32. doi: 10.1200/JCO.2016.67.0448. Epub 2016 Apr 4. PMID 27044935
- [Background] Catton CN, Lukka H, Gu CS, Martin JM, Supiot S, Chung PWM, Bauman GS, Bahary JP, Ahmed S, Cheung P, Tai KH, Wu JS, Parliament MB, Tsakiridis T, Corbett TB, Tang C, Dayes IS, Warde P, Craig TK, Julian JA, Levine MN. Randomized Trial of a Hypofractionated Radiation Regimen for the Treatment of Localized Prostate Cancer. J Clin Oncol. 2017 Jun 10;35(17):1884-1890. doi: 10.1200/JCO.2016.71.7397. Epub 2017 Mar 15. PMID 28296582
- [Background] Dearnaley D, Syndikus I, Mossop H, Khoo V, Birtle A, Bloomfield D, Graham J, Kirkbride P, Logue J, Malik Z, Money-Kyrle J, O'Sullivan JM, Panades M, Parker C, Patterson H, Scrase C, Staffurth J, Stockdale A, Tremlett J, Bidmead M, Mayles H, Naismith O, South C, Gao A, Cruickshank C, Hassan S, Pugh J, Griffin C, Hall E; CHHiP Investigators. Conventional versus hypofractionated high-dose intensity-modulated radiotherapy for prostate cancer: 5-year outcomes of the randomised, non-inferiority, phase 3 CHHiP trial. Lancet Oncol. 2016 Aug;17(8):1047-1060. doi: 10.1016/S1470-2045(16)30102-4. Epub 2016 Jun 20. PMID 27339115
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Michalski JM, Moughan J, Purdy J, Bosch W, Bruner DW, Bahary JP, Lau H, Duclos M, Parliament M, Morton G, Hamstra D, Seider M, Lock MI, Patel M, Gay H, Vigneault E, Winter K, Sandler H. Effect of Standard vs Dose-Escalated Radiation Therapy for Patients With Intermediate-Risk Prostate Cancer: The NRG Oncology RTOG 0126 Randomized Clinical Trial. JAMA Oncol. 2018 Jun 14;4(6):e180039. doi: 10.1001/jamaoncol.2018.0039. Epub 2018 Jun 14. PMID 29543933
- [Background] Kuban DA, Levy LB, Cheung MR, Lee AK, Choi S, Frank S, Pollack A. Long-term failure patterns and survival in a randomized dose-escalation trial for prostate cancer. Who dies of disease? Int J Radiat Oncol Biol Phys. 2011 Apr 1;79(5):1310-7. doi: 10.1016/j.ijrobp.2010.01.006. Epub 2010 May 20. PMID 20493642
- [Background] Dearnaley DP, Jovic G, Syndikus I, Khoo V, Cowan RA, Graham JD, Aird EG, Bottomley D, Huddart RA, Jose CC, Matthews JH, Millar JL, Murphy C, Russell JM, Scrase CD, Parmar MK, Sydes MR. Escalated-dose versus control-dose conformal radiotherapy for prostate cancer: long-term results from the MRC RT01 randomised controlled trial. Lancet Oncol. 2014 Apr;15(4):464-73. doi: 10.1016/S1470-2045(14)70040-3. Epub 2014 Feb 26. PMID 24581940
- [Derived] Fredman E, Icht O, Moore A, Bragilovski D, Kindler J, Golan S, Limon D. SABR-Dual: a phase II/III trial of two-fraction versus five-fraction stereotactic radiotherapy for localized low- and favorable intermediate-risk prostate cancer. BMC Cancer. 2024 Apr 8;24(1):431. doi: 10.1186/s12885-024-12165-1. PMID 38589860